CLINICAL TRIAL: NCT02466113
Title: A Multi-site, Open, Perspective Study of Prognostic Value and Benefit From Chemotherapy of Stage II Colon Cancer Based on a 6 microRNA Stratified Tool
Brief Title: A 6 microRNA Tool for Stratifying Stage II Colon Cancer of Receiving Adjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wu Song, Archiater, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015[28]
Record Dates: First submitted 2015-04-30; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Colonic Neoplasms; Effects of Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- An experimental group (Experimental): A 6 microRNA stratified tool is applied in this group.Investigators defined high risk patient and low risk patient according to the microRNA stratified tool.The high risk group should receive adjuvant chemotherapy while the low risk group observation.
  Interventions: Other: A 6 microRNA stratified tool
- A control group (Other): A classic stratified tool is applied in this group. Investigators defined high risk and low risk patient according to classical pathological features.The high risk group should receive adjuvant chemotherapy while the low risk group observation.
  Interventions: Other: A classic stratified tool

INTERVENTIONS:
Other: A 6 microRNA stratified tool — Investigators randomly assign patients to be assessed by a 6 microRNA stratified tool. MicroRNA(miRNA) tool contains miRNA of miR-21、miR-20a-5p、miR-103a-3p、miR-106b-5p、miR-143-5p and miR-215. Investigators evaluate these miRNA status of surgical specimens using qRT-PCR and calculate their risk score(risk score =(0.108×status of miRNA-21-5p)+(0.086×status of miRNA-20a-5p)+(0.240×status of miRNA-103a-3p)+(0.095×status of miRNA-106b-5p)-(0.238×status of miRNA-143-5p)-(0.237×status of miRNA-215),low expression status equals 0 and high expression status equals 1). Investigators defined high risk patient if their score larger than 1, the others as low risk patient.The high risk group should receive adjuvant chemotherapy while the low risk group deserve observation.
  Arms: An experimental group
Other: A classic stratified tool — Investigators randomly assign patients to be assessed by by classical pathological features. Pathological features include poorly differentiated histology(exclusive of those cancers that are MSI-H),lymphatic/vascular invasion,bowel obstruction and <12 lymph nodes examined. Investigators defined high risk patient if they had any pathological features, the others as low risk patient. The high risk group should receive adjuvant chemotherapy while the low risk group deserve observation.
  Arms: A control group

SUMMARY:
Whether patients with stage II colon cancer should receive adjuvant chemotherapy or not is still on debate.MicroRNA(miRNA) is a promising tool. Investigators invented a tool consisting of 6 miRNA(miR-21、miR-20a-5p、miR-103a-3p、miR-106b-5p、miR-143-5p and miR-215) that was effective to identify one should accept adjuvant chemotherapy or not. Here investigators randomly assign patients to be assessed by classical pathological features or the miRNA tool of determining who should accept chemotherapy. Disease free survival and overall survival are the end points of observation.

DETAILED DESCRIPTION:
Investigators randomly assign patients to be assessed by classical pathological features(control group) or the miRNA tool(experimental group). Pathological features include poorly differentiated histology(exclusive of those cancers that are MSI-H),lymphatic/vascular invasion,bowel obstruction and <12 lymph nodes examined.MicroRNA tool contains miRNA of miR-21、miR-20a-5p、miR-103a-3p、miR-106b-5p、miR-143-5p and miR-215. Investigators evaluate these miRNA status of surgical specimens using qRT-PCR and calculate their risk score(risk score =(0.108×status of miR-21-5p)+(0.086×status of miR-20a-5p)+(0.240×status of miR-103a-3p)+(0.095×status of miR-106b-5p)-(0.238×status of miR-143-5p)-(0.237×status of miR-215),low expression status equals 0 and high expression status equals 1). Investigators defined high risk patient if had any pathological features in control group or the score larger than 1 in the experimental group ,the others as low risk patient.The high risk group should receive adjuvant chemotherapy while the low risk group deserve observation. Primary endpoint is the disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed diagnosis of stage II colon cancer.
* With moderate/good ECOG health rating (PS): 0-1 score.
* The patient receive no anti-cancer treatment before primary surgery.
* The patient receive radical operation for colon cancer with negative margin.

Exclusion Criteria:

* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.
* Pregnant woman or lactating woman.
* With contraindication to receive adjuvant chemotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years or 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years or 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Song, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University